CLINICAL TRIAL: NCT01150929
Title: Rehabilitation After Total Knee Arthroplasty - Rotating Platform Versus Fixed Bearing Polyethylene
Brief Title: Rehabilitation After Total Knee Arthroplasty (TKA) - PFC Rotating Versus Fixed Bearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Silkeborg (Other); Gigtforeningen (Other); Protesekompagniet (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20050031
Record Dates: First submitted 2010-06-14; First posted 2010-06-25 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
Keywords: Knee arthroplasty; RSA; DXA; Gait analysis; Motion analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed bearing (Active Comparator): One of the 2 used implants.
  Interventions: Device: P.F.C. Sigma knee arthroplasty
- Rotating platform (Active Comparator): One of the 2 used implants.
  Interventions: Device: P.F.C. Sigma knee arthroplasty

INTERVENTIONS:
Device: P.F.C. Sigma knee arthroplasty — Randomization to either rotating platform or fixed bearing tibial plateau and polyethylene
  Other Names: PFC Sigma from DePuy International implants used.

SUMMARY:
The purpose of this study is to determine whether patient rehabilitation is equal for patients operated with two different knee implant designs.

The patients are randomized to treatment with either a simple hinge design implant (fixed bearing) or an implant with a mobile bearing polyethylene. This design difference might in principle enable the patients in the latter group to rehabilitate towards a more normal gait pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Silkeborg Regional Hospital, Orthopedic Dept. referred to total knee arthroplasty.

Exclusion Criteria:

* Neurologic disease with impact on gait.
* Orthopaedic disease ipsilateral hip joint.
* Patients outside the age limits.
* No informed consent signed.
* Patients suffering from dementia.
* Patients primarily included, but who perioperatively has their posterior cruciate ligament injured or sacrificed.
* Patients who later develop deep venous thrombosis or infection in the operated knee.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2012-08-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Radio Stereometric Analysis | 24 months
  Patients are analysed with stereo x-rays to asses implant micromigration.

SECONDARY OUTCOMES:
Gait analysis | 12 months
  Motion analysis is performed prior to surgery and after 6 and 12 months follow-up. Patients serve as their own control.
DXA | 24 months
  Dual Energy X-ray Absorptiometry (DXA) is used to asses bone mineral density (BMD) around the implant.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, DMsc, Study Chair — Aarhus Sygehus THG
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark